CLINICAL TRIAL: NCT02941835
Title: Preoperative Breast Irradiation, the PROBI Trial. A Phase I/II Feasibility Trial
Brief Title: Preoperative Breast Irradiation
Acronym: PROBI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow inclusion rate
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N16PRB; NL59561.031.16 (Registry Identifier: CCMO)
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: pre-operative radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- radiation (Other): intervention: pre-operative breast irradiation of 21 fx of 2.2Gy and boost 2.66Gy
  Interventions: Radiation: pre-operative irradiation

INTERVENTIONS:
Radiation: pre-operative irradiation — pre-operative whole breast irradiation of 21 fx of 2.2Gy and boost of 2.66Gy
  Other Names: radiotherapy

SUMMARY:
The PROBI is a phase I/II trial assessing the feasibility of preoperative whole breast irradiation in female patients with low to intermediate risk breast cancer, who undergo breast conserving therapy, including a boost dose of irradiation.

An additional goal of this study is to assess tumor response to radiotherapy, by imaging modalities (PET-CT and MRI) and pathology

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven invasive breast carcinoma
* cT1-2N0 breast cancer
* cM0
* female patients ≤ 50 years
* planned breast conserving surgery
* ability to undergo irradiation and surgery
* signed written informed consent

Exclusion Criteria:

* prior surgery or radiotherapy for the protocol tumor (neoadjuvant chemotherapy or endocrine therapy is allowed)
* planned oncoplastic reduction mammoplasty
* cTis
* extensive calcifications on mammagram (Birads 3,4 or 5)
* cT3-4 and/or cN1-3 invasive carcinoma
* distant metastasis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
Postoperative surgical complications | within six weeks after surgery
  postoperative complication will be scored by a specific list

SECONDARY OUTCOMES:
Radiological response | 6 weeks post-radiation
  assessed by MRI
Pathological response | at surgery
  surgery specimen
cosmetic outcome | 1,3 and 5 years post-treatment
  cosmesis will be scored by physician by questionnaire and cosmesis will be cored by patient by questionnaire

OTHER OUTCOMES:
gene expression profiles | 6 weeks
  at start a biopsy will be taken and compared to the surgical specimen at 6 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Scholten, MD, PhD, Principal Investigator — Antoni van Leeuwenhoek
Locations (1):
- Netherlands Cancer Institute, Amsterdam, Netherlands

REFERENCES:
- [Background] Bartelink H, Maingon P, Poortmans P, Weltens C, Fourquet A, Jager J, Schinagl D, Oei B, Rodenhuis C, Horiot JC, Struikmans H, Van Limbergen E, Kirova Y, Elkhuizen P, Bongartz R, Miralbell R, Morgan D, Dubois JB, Remouchamps V, Mirimanoff RO, Collette S, Collette L; European Organisation for Research and Treatment of Cancer Radiation Oncology and Breast Cancer Groups. Whole-breast irradiation with or without a boost for patients treated with breast-conserving surgery for early breast cancer: 20-year follow-up of a randomised phase 3 trial. Lancet Oncol. 2015 Jan;16(1):47-56. doi: 10.1016/S1470-2045(14)71156-8. Epub 2014 Dec 9. PMID 25500422
- [Background] Donker M, Straver ME, Wesseling J, Loo CE, Schot M, Drukker CA, van Tinteren H, Sonke GS, Rutgers EJ, Vrancken Peeters MJ. Marking axillary lymph nodes with radioactive iodine seeds for axillary staging after neoadjuvant systemic treatment in breast cancer patients: the MARI procedure. Ann Surg. 2015 Feb;261(2):378-82. doi: 10.1097/SLA.0000000000000558. PMID 24743607
- [Background] Egro FM, Pinell-White X, Hart AM, Losken A. The use of reduction mammaplasty with breast conservation therapy: an analysis of timing and outcomes. Plast Reconstr Surg. 2015 Jun;135(6):963e-971e. doi: 10.1097/PRS.0000000000001274. PMID 26017612
- [Background] Jones HA, Antonini N, Hart AA, Peterse JL, Horiot JC, Collin F, Poortmans PM, Oei SB, Collette L, Struikmans H, Van den Bogaert WF, Fourquet A, Jager JJ, Schinagl DA, Warlam-Rodenhuis CC, Bartelink H. Impact of pathological characteristics on local relapse after breast-conserving therapy: a subgroup analysis of the EORTC boost versus no boost trial. J Clin Oncol. 2009 Oct 20;27(30):4939-47. doi: 10.1200/JCO.2008.21.5764. Epub 2009 Aug 31. PMID 19720914
- [Background] van de Vijver MJ, He YD, van't Veer LJ, Dai H, Hart AA, Voskuil DW, Schreiber GJ, Peterse JL, Roberts C, Marton MJ, Parrish M, Atsma D, Witteveen A, Glas A, Delahaye L, van der Velde T, Bartelink H, Rodenhuis S, Rutgers ET, Friend SH, Bernards R. A gene-expression signature as a predictor of survival in breast cancer. N Engl J Med. 2002 Dec 19;347(25):1999-2009. doi: 10.1056/NEJMoa021967. PMID 12490681